CLINICAL TRIAL: NCT04841941
Title: A Feasibility Study to Assess the Visual Performance and Comfort of Hanita G4 Multifocal Soft Contact Lenses for Presbyopia at Normal Daily Routine Use.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: G4Multi
Record Dates: First submitted 2021-03-09; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): G4 Multifocal soft contact lens with a 54% water content for presbyopia
  Interventions: Device: G4 Multifocal soft contact lens with a 54% water content for presbyopia

INTERVENTIONS:
Device: G4 Multifocal soft contact lens with a 54% water content for presbyopia — The participants must agree to wear lenses from a trial set with the fit assessed according to the "Fitting Guide". Prescription lenses will then be ordered from the manufacturer.

SUMMARY:
The G4 Multi multifocal contact lens is a soft contact lens intended to correct far, intermediate, and near vision for individuals with presbyopia. The lens covers the cornea and part of the sclera. The lenses can be used for daily wear for up to 1 year.

DETAILED DESCRIPTION:
Study Design:

A clinical performance study without a control group to compare the G4Multi contact lens to other approved soft contact lenses for presbyopia

Study Objectives:

1. To assess the multifocal vision in the various ranges of the HANITA G4 Multi.
2. To rate the comfort of the lenses in individuals with presbyopia

Study population:

Healthy men and women above the age of 18 diagnosed with presbyopia who have used contact lenses in the past

Recruitment :

A total of 30 subjects completing at least 1 month of participation.

ELIGIBILITY:
Inclusion Criteria:

1. Presbyopia participants with healthy eyes who are not using any ocular medications, aged 18 years and over and who have used contact lenses in the past
2. Lens powers within the range available for the test lenses
3. Best spectacle-corrected visual acuity equal or greater than 20/25 (less than or equal to Log MAR 0.1)

Exclusion Criteria:

1. Anterior segment infection, inflammation, or abnormality
2. Any active anterior segment ocular disease that would contraindicate contact lens wear
3. The use of systemic or ocular medications that would contraindicate contact lens wear
4. History of herpetic keratitis
5. History of refractive surgery or irregular cornea
6. Slit lamp findings that are more serious than grade 1
7. Corneal vascularization greater than 1 mm of penetration
8. Pathologically dry eye;
9. Participation in a contact lens or contact lens care product clinical trial within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Assess visual acuity | 11-12 months
  Distance (far) manifest refraction and the testing distance used will be recorded on the case report forms. Manifest refraction will be determined using the maximum plus for best visual acuity method. The distance manifest refraction will be measured with a distance adjusted chart but not less than 4 meters. The actual manifest refraction distance will be noted on the case report forms.
  Results will be recorded in a Log Mar scale.

SECONDARY OUTCOMES:
Assess subjective degree of comfort while wearing the lenses | 11-12 months
  Participants will be asked to fill in a "Subjective Use Questionnaire" (appendix 2) .
SLIT LAMP EXAM | 11-12 months
  The slit lamp exam will include the entire cornea, sclera and conjunctiva exclusion symptoms:
  See ISO 11980 Annex B (informative) Procedures for the evaluation of safety, physiological performance and effects on ocular tissues.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - CLC, Raanana
  - Bar Ilan, Ramat Gan